CLINICAL TRIAL: NCT06384690
Title: Large-Scale, Sustainable, Nutrient-Dense MicroVeg: Generating Health Evidence & Production Capacity to Support Incorporation Into UK Diet
Brief Title: Generating Health Evidence From Dietary Supplementation With a Micro-vegetable Blend
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Advanced Growers Limited (Unknown); Ecog Pro Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 4331899
Record Dates: First submitted 2024-04-15; First posted 2024-04-25 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micro-vegetable blend (Experimental)
  Interventions: Dietary Supplement: Micro-vegetable blend
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Micro-vegetable blend — The intervention in this study is 6 weeks with a daily proprietary blend micro-vegetables that has been freeze-dried
  Arms: Micro-vegetable blend
Dietary Supplement: Placebo — The intervention in this study is 6 weeks with a placebo supplement
  Arms: Placebo

SUMMARY:
Micro-vegetables (MV) are seedlings of larger vegetables. They can be grown quickly and are a concentrated source of micronutrients. MV are thought to have broad health benefits, including many inflammatory conditions. These include metabolic, cardiovascular, and cognitive diseases. This could have important implications for the health of an ageing UK population. Less than a third of British adults consume 5 portions of fruit and vegetables per day; this is the level that reduces risk of morbidity and mortality. Vegetables, including MV may - at least in part - exert their health effects by changing the level and type of bacteria in the mouth and gut. Despite their promise, the MV scientific literature is not yet extensive enough to support definitive health claims. It requires the addition of high-quality studies that are relevant to humans. This study will firstly investigate the anti-inflammatory effects on skeletal muscle and adipose tissue in older adults, using a proteomics approach. Second, this study will assess concentrations of circulating inflammatory markers in the sera collected from participants at baseline and at the conclusion of a 6-week period. Further, this study will describe the effects of six weeks MV consumption on cognition, and the oral and gut microbiome. As the bioactive compounds in the MV are owed to the potential beneficial effects for human health, these will be characterised in sera collected from participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years and above
* Body mass index > 25kg/m2
* Able to give written informed consent to participate in the study

Exclusion Criteria:

* Not meeting any inclusion criteria
* Have had an adverse reaction to a local anaesthetic in the past
* Hepatitis B, Hepatitis C or HIV positive
* Have a bleeding disorder or are regularly taking a medication that will impair their blood's capacity to clot (e.g., aspirin, clopidogrel, warfarin, heparin)
* Have had a severe adverse reaction to plasters
* Have a gastrointestinal disorder that may impair the absorption of the supplement from the gastrointestinal tract
* Have an autoimmune condition
* Have a diagnosed neurocognitive disorder
* Have a skin condition that is likely to increase the risk of infection at the biopsy site
* Frequent use of medication or recreational drugs likely to affect our results
* Recent infection or vaccination
* Known allergy to any vegetables
* Participated in a nutrition supplementation study in the last month

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Tandem Mass Tag (TMT) global proteomics | Adipose and skeletal muscle sampling at baseline and 6-week post-intervention
  Characterisation of the proteome - hypothesis free

SECONDARY OUTCOMES:
Concentration of broad panel of inflammatory cytokines | Blood sample collected at baseline and 6-week post-intervention
  Using multiplex immunoassay including but not limited to TNFα, IL-6, IL-10 and IL-1β, MIP1α, Galectin 1, Chemerin, Eotaxin, gp130, MCP-1, IL-7, MIP3α, IL-15, Aggrecan, Resistin, Leptin, MIP1β, MMP-1, MMP-3, MMP-13, and FABP4
Concentration of circulating bioactive components | Blood sample collected at baseline and 6-week post-intervention
  Characterisation of bioactive components, including but not limited to polyphenols
Microbiome | Faecal and saliva collected at baseline and 6-week post-intervention
  Metagenomic sequencing. Exploratory outcome to establish reference data for Shannon H diversity index and Chao1 species richness
Simple Reaction Time | 5 times throughout the intervention (baseline, week 2, week 4, week 6 and week 8)
  Assessment of alertness and focused attention
Digit Vigilance | 5 times throughout the intervention (baseline, week 2, week 4, week 6 and week 8)
  Assessment of sustained and intensive attention
Choice Reaction Time | 5 times throughout the intervention (baseline, week 2, week 4, week 6 and week 8)
  Accompanied with Simple Reaction Time and records additional time taken to execute appropriate response
Pattern Separation | 5 times throughout the intervention (baseline, week 2, week 4, week 6 and week 8)
  Assessment of ability to store and retrieve visual information

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health and Sports Sciences, University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No